CLINICAL TRIAL: NCT06221046
Title: Prospective Evaluation of the Safety and Efficacy of an Enhanced Barrier Cream for the Treatment of Moisture Associated Skin Damage
Brief Title: Testing the Safety and Efficacy of a Novel Barrier Cream for the Treatment of Moisture Associated Skin Damage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scotiaderm (Other)
Collaborators: The Salvation Army Toronto Grace Health Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-DRM-001
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Moisture Associated Skin Damage; Incontinence Associated Dermatitis; Fecal Incontinence
Keywords: MASD; Moisture Associated Skin Damage; Incontinence Associated Dermatitis; IAD; Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, double-blind, controlled study. This study will follow 60 patients in medical units at Toronto Grace Health Centre who present with IAD from diarrhea and/or fecal incontinence. Randomizations will be done by medical unit. Patients will be enrolled in each participating unit until 30 patients are recruited in each study arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomizations will be performed by unit, such that each participating unit provides the same treatment to all patients within that unit. This minimizes error in the supply chain of study product. The research coordinator will have a list of the randomizations; this will not be shared with the investigator, the care team, or the participants. Study product will be provided in identical, plain white tubes with labels separate in the shipping container. The study coordinator will ensure that each participating unit receives the correct product (study intervention or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients in units randomized to the control arm will be treated with a zinc oxide barrier cream, which is standard of care for MASD.
  Interventions: Drug: Control (Standard treatment)
- Investigational Product (Experimental): Patients in units randomized to the intervention arm will be treated with Scotiaderm's novel barrier cream, Dermategrity "anti-fecal" barrier cream.
  Interventions: Other: Novel Barrier Cream

INTERVENTIONS:
Drug: Control (Standard treatment) — Patients in the control arm will be treated with a standard zinc oxide barrier cream. Scotiaderm will supply the control product, such that the formula is identical to the intervention with the only difference being the addition of plant extract in the investigational product.
  Other Names: Zinc Oxide Barrier Cream
  Arms: Control
Other: Novel Barrier Cream — Patients randomized to the intervention arm will receive treatment with Scotiaderm's proprietary barrier cream formula. This product contains soy extract for enhanced healing of MASD secondary to fecal incontinence.
  Other Names: Dermategrity "Anti-fecal" Barrier Cream
  Arms: Investigational Product

SUMMARY:
Liquid stool and diarrhea are associated with an increased risk for moisture-associated skin damage (MASD), and clinical evidence suggests that exposure to liquid stool is associated with severe MASD and extensive erosion of affected skin. There are no known products on the market that treat fecal incontinence or MASD caused by fecal enzyme activity.

Scotiaderm has invented a novel barrier cream (Dermategrity "Anti-fecal" Barrier Cream) with an enhanced formula containing zinc oxide and soybean extract that inhibits fecal enzymes to protect the skin while preventing further breakdown. Dermategrity "Anti-fecal" Barrier Cream has shown superior outcomes in comparison to zinc oxide alone in simulated laboratory testing, and promising results have been obtained in clinical case studies. To date, however, there has been no formal clinical testing of this new barrier product in comparison to standard zinc oxide creams.

The purpose of this study is to perform a randomized, controlled clinical study comparing Dermategrity "Anti-fecal" Barrier Cream to zinc oxide barrier cream to determine if there is a difference in healing, clinical outcomes, and the speed of resolution of MASD symptoms between groups.

DETAILED DESCRIPTION:
Moisture associated skin damage (MASD) is a grouping of painful, irritating rashes which occur when a patient has repeated or prolonged exposure to moisture from perspiration, urine and/or feces. Commonly encountered rashes in this group include incontinence-associated dermatitis (IAD) and intertrigo (ITD). These conditions can affect as many as one in five hospitalized patients and up to 50% of intensive care unit patients, putting them at risk of skin breakdown, serious infection, and the development of pressure ulcers. MASD is a common but overlooked and under-reported skin care problem, and there are many gaps in the knowledge of how best to treat these rashes.

Liquid stool and diarrhea are associated with an increased risk for MASD when fecal materials remain in contact with the skin for a prolonged period. Diarrhea is associated with an increased likelihood of IAD in children, and clinical evidence suggests that exposure to liquid stool is associated with severe MASD and extensive erosion of affected skin. Liquid stool is also rich with coliform bacteria, and the gastrointestinal tract acts as a reservoir for various fungal species including Candida, which commonly complicates IAD. Liquid stool contains higher concentrations of proteolytic enzymes with the potential to impair the moisturizing effects of proteins such as filaggrin, and the softening effects of the intrinsic lipids in the skin, both of which are vital in maintaining the barrier functions in skin. These effects are exacerbated by a more alkaline pH and the higher concentrations of active fecal enzymes associated with diarrhea. Research on incontinent patients in the intensive care unit shows that the mean time to development of MASD is 4 days. The presence of liquid stool is an independent risk factor for the development of IAD, with patients developing IAD at a rate of 1.5x that of patients who are continent.

The current standard of care for the treatment and prevention of MASD involves a structured skin care regiment that involves cleansing of the skin to remove excessive moisture and irritants with a pH balanced cleanser, moisturizing the skin when indicated and applying a protective productive product when repeated exposure to moisture is anticipated. There are many factors that influence the choice of moisturizers and protective products, however a Cochrane review of IAD in 2016 noted that there was no evidence that one product was superior to another. Currently, a single-step intervention using disposable washcloths that incorporate cleansing, protecting, and skin restoring agents into a single product (3-in-1 wipes) is widely practiced and helps to maximize adherence to best practices in the treatment and prevention of MASD.

Research has shown that a family of enzyme inhibitors can be isolated from a subset of plants. These plant-based inhibitor peptides (PBIPs) have been well characterized and have been shown to reduce the proteolytic activities of enzymes commonly seen in the digestive tract and feces. PBIPs have demonstrated anticarcinogenic activity against tumor cells in vitro, in animal models, and in human phase II clinical trials. PBIP Concentrates (PBIPCs) have the same anticarcinogenic profile as purified PBIPs and have been developed for human trials. Both PBIPs and PBIPCs are nontoxic, and safety has been reported in numerous clinical studies. Topical PBIPCs have been used safely in clinical studies as hair growth suppressant and to treat skin pigmentation.

Scotiaderm Inc. has developed Dermategrity "Anti-fecal" Barrier Cream; a topical formulation of a barrier cream containing zinc oxide with PBIPCs from soybeans to be used in the treatment of MASD caused by diarrhea and/or fecal incontinence. The purpose of the proposed research is to explore the safety and efficacy of soy extract incorporated into a standard barrier in the treatment of MASD from diarrhea or fecal incontinence. The goal of this research is to conduct a randomized, double-blind, controlled study in inpatients in medical care units who present with diarrhea and/or fecal incontinence.

This is a single center, randomized, double-blind, controlled study of 60 patients. Patients will be treated with barrier cream daily, with an application after each bowel movement. There is no maximum number of applications, however patients must be given a minimum of two applications/day to adequately protect the skin. Patients will be followed for two weeks, with a baseline/enrollment visit, daily visits for the first week of participation, and a final visit on day fourteen. For the first week of the study, the principal investigator or designated study staff patients will complete a daily assessment of the patient's rash, including the Global IAD assessment, an image of the rash, and the VAS erythema score. TEWL and colorimeter measurements, as well as adverse event reporting, will also be completed daily for the first week. For the second week of study participation, cream application will follow the same protocol, however daily assessments will not occur.

The clinical care team providing treatment to the patients will be blinded to their group assignment. The research coordinator will provide the clinical team with a plain tube of barrier cream and an envelope outlining the treatment protocol for the study arm the patient has been assigned. The study product will be shipped with the product labels included and these labels will be kept on file by the study coordinator for reference as needed. For all applications, a qualified healthcare professional (nurse, physician, physician assistant, etc.) will apply the treatment to the patient.

At baseline, demographic information will be collected. A qualified member of the study team (PI, research nurse, etc.) will complete the daily clinical assessments using the Global IAD and the CAN MASD. Photographs, the VAS Erythema score, TEWL and colorimeter measurements, and case report forms will be completed by a designated member of the study team. For all images which are collected in the study, identifying features such as tattoos and birthmarks that are unavoidable to capture will be blurred on the stored images. When collecting images of incontinence-associated rashes genitalia cannot be avoided in all instances, however, in any instance in which the genitalia is not encompassed by the rash, it will not be included in the digital image.

After capturing images from the region of concern the healthcare provider will clean the area with 3-in-1 perineal wipes and allow the skin to air dry for five minutes. The treatment (either experimental or control arm cream) will be applied according to the provided instructions for use a minimum of two times per day or following each episode of incontinence for each of the fourteen days of study enrollment.

Follow-up Assessments:

For all remaining days of study, the protocol will be as follows: the standard measurement scale and red adhesive label will be applied, and an image of the rash will be taken. No identifying features will be included. The rash will be treated with the arm 1 or arm 2 protocol for seven days. After completion of the study, the container which housed the cream will be weighed and the total weight of cream used will be recorded.

The clinical care team providing treatment to the patients will be blinded to their group assignment. The research coordinator will provide the clinical team with a plain tube of barrier cream and an envelope outlining the treatment protocol for the study arm the patient has been assigned. The study product will be shipped with the product labels included and these labels will be kept on file by the study coordinator for reference as needed. For all applications, a qualified healthcare professional (nurse, physician, physician assistant, etc.) will apply the treatment to the patient.

At baseline, demographic information will be collected. A qualified member of the study team (PI, research nurse, etc.) will complete the daily clinical assessments using the Global IAD and the CAN MASD. Photographs, the VAS Erythema score, TEWL and colorimeter measurements, and case report forms will be completed by a designated member of the study team. For all images which are collected in the study, identifying features such as tattoos and birthmarks that are unavoidable to capture will be blurred on the stored images. When collecting images of incontinence-associated rashes genitalia cannot be avoided in all instances, however, in any instance in which the genitalia is not encompassed by the rash, it will not be included in the digital image.

After capturing images from the region of concern the healthcare provider will clean the area with 3-in-1 perineal wipes and allow the skin to air dry for five minutes. The treatment (either experimental or control arm cream) will be applied according to the provided instructions for use a minimum of two times per day or following each episode of incontinence for each of the fourteen days of study enrolment.

For all remaining days of study, the protocol will be as follows: the standard measurement scale and red adhesive label will be applied, and an image of the rash will be taken. No identifying features will be included. The rash will be treated with the arm 1 or arm 2 protocol for seven days. After completion of the study, the container which housed the cream will be weighed and the total weight of cream used will be recorded.

Due to the novelty of the product and the limited number of clinical research studies on MASD, there is no existing data with which to base a sample size calculation on. Consequently, the study proposes to enroll 60 patients (30/group), as 30 samples is considered the minimum sufficient number to achieve a normal distribution. Data from the first 20-30 patients enrolled in the study will be used as pilot data to perform a power analysis, and if adjustments are required to adequately power the study (either more or less participants needed), an amendment request will be made.

The primary analysis will focus on the safety and efficacy of the active agent in Dermategrity "Anti-fecal" Barrier Cream in the treatment of MASD associated with diarrhea and/or fecal incontinence. Safety will be assessed by documenting any adverse events/reactions that occur to patients while participating in this study. Efficacy will be assessed by quantifying the change in VAS Erythema score from day 0 to day 7 and day 14. A repeated measures ANOVA will be used to compare outcomes across time points for each of the independent variables. For categorical data, frequencies and percentages will be provided. For continuous data, descriptive statistics, including sample size, mean, median, standard deviation, and range of values (minimum and maximum) will be provided. A significance level of alpha = 0.05 will be used for all statistical tests and a p-value < 0.05 will be considered statistically significant unless otherwise specified. 95% confidence intervals will be presented whenever appropriate.

We hypothesize that a barrier cream containing soy extract will demonstrate an excellent safety profile and accelerate healing of MASD due to diarrhea and/or fecal incontinence compared to the standard of care (zinc oxide barrier cream) over a two-week period.

ELIGIBILITY:
Patients who meet all the below criteria will be eligible for inclusion in the study:

* ≥18 years of age;
* Clinical diagnosis of incontinence-associated dermatitis resulting from diarrhea and/or fecal incontinence;
* Minimum expected stay in hospital of two weeks;
* Able to provide written informed consent (OR consent by a recognized substitute-decision maker) including explicit consent to take daily photographs of the rash associated with MASD.

Patients who meet any of the following exclusion criteria will not be eligible for enrolment:

* History of complex skin disorders (such as psoriasis or eczema);
* Allergy to any of the ingredients in the study product;
* Visual evidence of a bacterial skin infection;
* Anticipated length of stay in hospital less than two weeks;
* Life expectancy less than two weeks;
* Use of a dressing or bandage covering the rash that cannot reasonably be removed for required study activities without compromising patient comfort or care.

Note: Patients who are pregnant will not be excluded from the study unless they present with a rash or other skin conditions that may confound assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
GLOB-IAD Clinical Assessment | 14 days
  The GLOB-IAD Clinical Assessment is the only validated clinical tool for assessing MASD. This assessment will be performed daily for the first 7 days, and once again at day 14. All GLOB-IAD assessments will be done by a qualified study team member (i.e., principle investigator, wound care nurse, etc.).
Visual Analog Scale for Erythema | 14 days
  The Visual Analog Scale (VAS) for erythema is a visual assessment tool to measure the severity of a patient's erythema. The VAS Erythema employs a visual scale from "no visible signs of erythema" to "worst possible erythema", allowing the investigator to capture erythema for all skin colors and types. The VAS Erythema will be performed daily for 7 days, and once again on day 14.
Safety - Adverse Events and Product-Related Adverse Effects | 14 days
  Safety of the investigational product will be assessed by documenting the frequency and severity of adverse events, and their relationship to the investigational product.

SECONDARY OUTCOMES:
Trans-epidermal Water Loss (TEWL) | 14 days
  Increased loss of water through the epidermis is indicitive of reduced integrity of the skin;s natural barrier. Trans-epidermal water loss from the area affected by MASD will be measured using a TEWL probe (Tewameter TM Hex Probe). TEWL will be measured daily for 7 days, and once again on day 14.
CAN MASD Assessment Tool | 14 days
  The CAN MASD is a novel assessment tool for MASD. This study will test the reliability and validity of the CAN MASD for assessing MASD in a clinical setting, compared to the only other validated assessment tool for IAD, the GLOB-IAD. CAN MASD Assessments will be performed daily for 7 days, and once again on day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Woo, PhD, RN, NSWOC WOCC(C), Principal Investigator — Toronto Grace Health Centre

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.